CLINICAL TRIAL: NCT03916757
Title: Open-label Phase II Trial of the Safety and Efficacy of V-Boost in Patients With Refractory Glioblastoma Multiforme (GBM)
Brief Title: V-Boost Immunotherapy in Glioblastoma Multiforme Brain Cancer
Acronym: GBM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Imm008
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme; Glioma of Brain
Keywords: Brain cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients who passed eligibility requirement will receive daily dose of V-Boost
Masking Description: This is open label study, no masking is required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-Boost recipients (Experimental): In this open label study all eligible participants will receive daily tablet of V-Boost
  Interventions: Biological: V-Boost

INTERVENTIONS:
Biological: V-Boost — Open label setting
  Other Names: V-Boost Immunitor

SUMMARY:
The Phase II study to determine the safety and efficacy of V-Boost in treating a type of brain cancer called Glioblastoma Multiforme (GBM). V-Boost is an immunotherapy in which the patient's immune system will be modulated to eliminate tumor cells. V-Boost is made as an oral tablet which contains specially formulated hydrolyzed GBM antigens along with alloantigens. Patients are either newly diagnosed or with recurrent form of GBM who may have been subjected to surgery and/or chemo- or radiation therapy that ended up unsuccessful. The goal is to eradicate GBM tumor cells through daily oral administration of one pill of V-Boost immunotherapeutic vaccine, which so far has not shown any adverse reaction.

DETAILED DESCRIPTION:
The proposed Phase II trial is an-open label study of the safety and efficacy of V-Boost in newly diagnosed or treatment-refractory patients with glioblastoma multiforme (GBM) following unsuccesfull resection and/or chemoradiation. The Phase I clinical tria,l carried out in a small, open-label study, demonstrated safety and promising efficacy. The purpose of this study is to gain additional information from a larger clinical trial aimed to recruit at least 20 patients with GBM. Patients may be newly diagnosed with GBM or are those who have been subjected to resection and/or chemotherapy or radiation, but without success. Patients need to have imaging records and health assessment prior to study enrollment. Those on chemotherapy or radiation can be in washout period or may receive immunotherapy concurrently. Patients will be administered daily dose of V-Boost oral tablet for at least one month and additional dosing can be envisaged depending on outcome of first month. The primary objective is to evaluate the effect on tumor size and progression free survival (PFS) in comparison to patients on standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of GBM
* ≥ 5 years of age
* Consent from parents or legal guardian if under-aged

Exclusion Criteria:

* Severe pulmonary, cardiac or other systemic disease
* Presence of an acute infection requiring active treatment with antibiotics/antivirals
* Receiving corticosteroids (e.g., dexamethasone) during study duration

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Effect on tumor size | 3 months
  Imaging of brain at 3-month time post-therapy and comparison to baseline records

SECONDARY OUTCOMES:
Effect on progression-free survival | 3 months
  Evaluation of patients status on progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbayar, MD/PhD, Study Chair — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

REFERENCES:
- [Background] Tarakanovskaya MG, Chinburen J, Batchuluun P, Munkhzaya C, Purevsuren G, Dandii D, Hulan T, Oyungerel D, Kutsyna GA, Reid AA, Borisova V, Bain AI, Jirathitikal V, Bourinbaiar AS. Open-label Phase II clinical trial in 75 patients with advanced hepatocellular carcinoma receiving daily dose of tableted liver cancer vaccine, hepcortespenlisimut-L. J Hepatocell Carcinoma. 2017 Apr 12;4:59-69. doi: 10.2147/JHC.S122507. eCollection 2017. PMID 28443252
- See also: link to similar study — https://www.ncbi.nlm.nih.gov/pubmed/28443252